CLINICAL TRIAL: NCT03772288
Title: A Phase 1b Study of TAK-659 in Combination With NKTR-214 in Patients With Advanced Non-Hodgkin Lymphoma
Brief Title: A Study of TAK-659 in Combination With NKTR-214 in Participants With Advanced Non-Hodgkin Lymphoma (NHL)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Decision: No Safety or Efficacy Concerns
Sponsor: Calithera Biosciences, Inc (Industry)
Collaborators: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C34015; U1111-1218-4372 (Registry Identifier: WHO)
Record Dates: First submitted 2018-12-10; First posted 2018-12-11 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Drug Therapy
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — TAK-659; bempegaldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation: TAK-659 + NKTR-214 (Experimental): TAK-659 tablet, orally, once daily along with NKTR-214, infusion, intravenously, once on Day 1 in a 21-day treatment cycle, until disease progression, unacceptable toxicities, or discontinuation by participant. The dose escalation phase will determine the MTD or RP2D of TAK-659. Dose escalation of TAK-659 will be based on available safety and tolerability data.
  Interventions: Drug: TAK-659; Drug: NKTR-214
- Safety Expansion: TAK-659 + NKTR-214 (Experimental): TAK-659, tablet, orally, once daily along with NKTR-214, infusion, intravenously, once on Day 1 of 21-day treatment cycle, until disease progression, unacceptable toxicities, or discontinuation by participants. TAK-659 and NKTR-214 MTD/RP2D will be determined from the dose escalation phase.
  Interventions: Drug: TAK-659; Drug: NKTR-214

INTERVENTIONS:
Drug: TAK-659 — Tablets.
Drug: NKTR-214 — Intravenous infusion.

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) for TAK-659 when administered in combination with NKTR-214.

DETAILED DESCRIPTION:
The drugs that are being tested in this study are TAK-659 and NKTR-214. TAK-659 in combination with NKTR-214 is being tested for participants with advanced B-cell NHL, including DLBCL, FL, MZL, or MCL, after 2 prior lines of therapy. The study will determine the MTD or the RP2D of TAK-659 when administered with NKTR-214.

The study will enroll approximately 40 participants, approximately 18 to 24 participants in a dose escalation phase, and approximately 12 participants will be added after determination of MTD/RP2D in the safety expansion phase. This study consists of 2 phases: a dose escalation phase and a safety expansion phase.

TAK-659 and NKTR-214 doses will be escalated according to a modified 3+3 dose escalation schema. TAK-659 60 milligram (mg) + NKTR-214 0.003 milligram per kilogram (mg/kg) is the starting dose. Participants could also receive 80 mg once daily (QD) TAK-659 during dose escalation and 0.003mg/kg or 0.006mg/kg of NKTR-214. Lower doses (example 40 mg) and/or alternative regimens (including intermittent dosing) or schedules of TAK-659 are permissible following discussion between sponsor and investigators. In dose escalation phase, dose levels will be escalated based on available safety and tolerability data to determine the MTD or RP2D. Dose for safety expansion phase will be based on available safety, pharmacodynamics, and preliminary efficacy data.

For participants enrolled in either the dose escalation or safety expansion phases, the maximum duration of treatment will be 12 months unless, in the opinion of the investigator and with the agreement of the sponsor, the participant would derive benefit from continued therapy beyond 12 months. Participants will make multiple visits to the clinic, and will have an end of treatment visit 30 days after the last dose of TAK-659 or NKTR-214 or before the start of subsequent alternative anticancer therapy, whichever occurs first. Participants will be followed for 90 days after the last dose or subsequent anti-cancer therapy, whichever occurs first, to permit the detection of any delayed treatment-related adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of advanced B-cell NHL, including diffuse large B-cell lymphoma (DLBCL), follicular lymphoma (FL), marginal zone lymphoma (MZL), or mantle cell lymphoma (MCL) (Waldenstrom macroglobulinemia [WM] and chronic lymphocytic leukemia [CLL]/small lymphocytic leukemia [SLL] are excluded).
2. Radiographically or clinically measurable disease with at least 1 target lesion per (greater than [>] 1.5 centimeter [cm] in the longest diameter for a lymph node or nodal mass, or >1.0 cm in the longest diameter for extranodal disease) Lugano 2014 criteria for malignant lymphoma.
3. Participants who are refractory or relapsed after at least 2 prior lines of therapy due to progression, intolerance, or physician/participant decision, and for whom no effective standard therapy is available per the investigator's assessment. The sponsor may restrict prior lines of therapy in the expansion phase of the study based on emerging data. The decision may be documented and shared with investigators in a memo before the initiation of the dose expansion phase followed by updating the exclusion criteria in a subsequent amendment, if deemed necessary. Requirements for prior therapy depending on disease type are outlined in the protocol, however all patients must be ineligible for or have already failed hematopoietic stem cell transplant.
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1 and life expectancy of >3 months.
5. Must have adequate organ function.
6. Recovered (that is, less than or equal to [<=] Grade 1 toxicity) from the clinically significant reversible effects of prior anticancer therapy.

Exclusion Criteria:

1. Central nervous system (CNS) lymphoma; active brain or leptomeningeal metastases, as indicated by positive cytology from lumbar puncture or computed tomography (CT) scan/magnetic resonance imaging. Exceptions include those participants who have completed definitive therapy, are not on steroids, have a stable neurologic status for at least 2 weeks after completion of the definitive therapy and steroids, and do not have neurologic dysfunction that would confound the evaluation of neurologic and other AEs.
2. Known human immunodeficiency virus (HIV) infection or HIV-related malignancy, hepatitis B surface antigen positive, or known or suspected active hepatitis C infection.
3. History of drug-induced pneumonitis requiring treatment with steroids; history of idiopathic pulmonary fibrosis, organizing pneumonia, or evidence of active pneumonitis on screening chest CT scan; history of radiation pneumonitis in the radiation field (fibrosis) is permitted.
4. Systemic anticancer treatment (including investigational agents) or radiotherapy less than 2 weeks before the first dose of study treatment (<=4 weeks for antibody-based therapy including unconjugated antibody, antibody-drug conjugate, and bi-specific T-cell engager agents; <=8 weeks for cell-based therapy or antitumor vaccine).
5. Participants in need of immediate cytoreductive therapy.
6. Prior autologous stem cell transplant (ASCT) within 6 months or prior ASCT at any time without full hematopoietic recovery, defined by the entry criteria in the study, before Cycle 1 Day 1 or allogeneic stem cell transplant any time.
7. Use or consumption of:

   * Medications or supplements that are known to be inhibitors of P-glycoprotein (P-gp) and/or strong reversible inhibitors of cytochrome (CYP3A), strong CYP3A mechanism-based inhibitors, strong CYP3A inducers or P-gp inducers within 5 times the inhibitor half-life or within 7 days before the first dose of study drug. In general, the use of these agents is not permitted during the study except in cases in which an AE must be managed.
   * Grapefruit-containing food or beverages within 5 days before the first dose of study drug. Note that grapefruit-containing food and beverages are not permitted during the study.
8. Active, known, or suspected autoimmune disease. Participants requiring systemic treatment within the past 3 months or with a documented history of clinically severe autoimmune disease that requires systemic steroids or immunosuppressive agents. (Exceptions include any patient taking 10 mg or less of prednisone or equivalent, participants with vitiligo, hypothyroidism stable on hormone replacement, type 1 diabetes, Graves disease, Hashimoto disease, alopecia areata, eczema, or with medical monitor approval.)
9. History of organ or tissue transplant that requires systemic use of immunosuppressive agents.
10. Prior treatment with TAK-659 or any spleen tyrosine kinase (SYK) inhibitor or interleukin-2 (IL-2) therapy.
11. Use of >2 antihypertensive medications for management of hypertension (including diuretics).
12. Major surgery within 14 days before the first dose of study drug and not recovered fully from any complications from surgery or systemic infection requiring intravenous antibiotic therapy or other serious infection within 14 days before the first dose of study drug.
13. Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of TAK-659, including difficulty swallowing tablets or diarrhea Grade >1 despite supportive therapy.
14. Treatment with high-dose corticosteroids for anticancer purposes within 14 days before the first dose of TAK-659; daily dose equivalent to 10 mg oral prednisone or less is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2021-11-10 (Estimated); Study Completion 2021-11-17 (Estimated)

PRIMARY OUTCOMES:
MTD of TAK-659 in Combination with NKTR-214 | 3 weeks after last dose of last participant in dose escalation or up to 6 months
RP2D of TAK-659 in Combination with NKTR-214 | 3 weeks after last dose of last participant in dose escalation or up to 6 months

SECONDARY OUTCOMES:
Cmax: Maximum Observed Plasma Concentration for TAK-659 | Cycle 1 and Cycle 2: Day 1 pre-dose and at multiple time points (up to 24 hours) post-dose (cycle length=21 days)
Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-659 | Cycle 1 and Cycle 2: Day 1 pre-dose and at multiple time points (up to 24 hours) post-dose (cycle length=21 days)
AUCτ: Area Under the Plasma Concentration-time Curve From Time During the Dosing Interval for TAK-659 | Cycle 1 and Cycle 2: Day 1 pre-dose and at multiple time points (up to 24 hours) post-dose (cycle length=21 days)
Cmax: Maximum Observed Plasma Concentration for NKTR-214 | Cycle 1 Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose (cycle length=21 days)
Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for NKTR-214 | Cycle 1 Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose (cycle length=21 days)
AUC: Area Under the Plasma Concentration-time Curve for NKTR-214 | Cycle 1 Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose (cycle length=21 days)
Overall Response Rate (ORR) | Through study completion, approximately 40 months
  ORR is defined as the percentage of participants in the response-evaluable population who achieved either complete response (CR) or partial response (PR) as assessed by the investigator according to the Lugano 2014 criteria.
Duration of Response (DOR) | From first CR or PR to progressive disease (PD) or relapse (through study completion, approximately 40 months)
  DOR is defined as the time from first CR or PR to PD or relapse in the response-evaluable population.
Progression-free Survival (PFS) | From first dose of study drug to PD or death (through study completion, approximately 40 months)
  PFS is defined as the time from first dose to PD or death in the response-evaluable population.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Millennium Pharmaceuticals, Inc.
Locations (6):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Henry Ford Hospital, Detroit, Michigan
  - New York University Langone Medical Center, New York, New York
- Canada (3):
  - Alberta Health Services, Calgary, Alberta
  - Jewish General Hospital, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke (CIUSSS de lEstrie - CHUS), Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.